CLINICAL TRIAL: NCT02693353
Title: Association of Cystoid Macular Edema After Cataract Surgery in Patients With and Without Epiretinal Membrane
Brief Title: Epiretinal Membrane and Pseudophakic Cystoid Macular Edema
Status: Terminated | Type: Observational
Why Stopped: Recent publication makes current study obsolete.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Sierpina, MD, Loma Linda University
Other Study IDs: 5150420
Record Dates: First submitted 2016-02-24; First posted 2016-02-26 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Macular Edema; Epiretinal Membrane
MeSH Terms: conditions — Macular Edema; Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study Group: Patients with diagnosed epiretinal membrane undergoing cataract surgery.
- Control Group: Patients without epiretinal membrane undergoing cataract surgery.

SUMMARY:
Prospective, observational cohort study evaluating the association between pre-surgical existence of an epiretinal membrane (ERM) and the development of pseudophakic cystoid macular edema (PCME) using spectral domain optical coherence tomography (OCT) measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Cataract surgery patients

Exclusion Criteria:

* Pre-existing macular edema
* Choroidal neovascularization
* Uveitis
* Age-related macular degeneration
* Myopia > 6 diopters
* Proliferative diabetic retinopathy
* Diabetics retinopathy great than mild in serverity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 who are undergoing cataract surgery at Loma Linda University Eye Institute
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cystoid Macular Edema diagnosed by OCT | Within 90 days post op

CONTACTS AND LOCATIONS:
Overall Officials: David Sierpina, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided